CLINICAL TRIAL: NCT05039957
Title: Management of Fracture Ankle in Patients With Uncontrolled Diabetes by Hind Foot Nail With Versus Without Joint Preparation: Randomized Control Study
Brief Title: Management of Fracture Ankle in Adults With Uncontrolled Diabetes by Hind Foot Nail With Versus Without Joint Preparation , in Assiut University Hospital
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, momen ayman fekry, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17200615
Record Dates: First submitted 2021-09-02; First posted 2021-09-10 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Figure Out the Best Method of Fixation for Management of Patients With Diabetic Fracture Ankle

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Active Comparator)
  Interventions: Other: joint preparation
- B (Experimental)
  Interventions: Other: without joint preparation

INTERVENTIONS:
Other: joint preparation — fixation of fracture with joint preparation
  Arms: A
Other: without joint preparation — fixation of fracture without joint preparation
  Arms: B

SUMMARY:
Diabetes is a well-known risk factor for complications following ankle fracture fixation.Current recommendations for operative treatment of ankle fractures in patients with diabetes consist of increased rigid fixation and prolonged periods of non-weight bearing with minimally invasive techniques.

Yee et al described a treatment algorithm for ankle fractures in diabetes patients based on the extent of their diabetic complications, Adelaide Fracture in the Diabetic Ankle (AFDA) score, and suggest that primary ankle arthrodesis may be an option in severe situations.

Ebaugh et.al. described the technique of fixing the ankle joint in diabetic patients without joint preparation .

Primary hindfoot arthrodesis with Calcaneotibial nail with formal joint preparation was described by many authors as treatment for ankle fractures in diabetic patient .

To our knowledge, there is no comparative study in management of ankle fractures in diabetic patients using these two different techniques.

Our hypothesis is to try to prove that management of diabetic fracture ankle by hindfoot nail without joint preparation is better than other techniques regarding overall lower complication rate, higher functional outcome and better option for treatment of these patients using minimal invasive approaches in those high risk patients.

ELIGIBILITY:
Inclusion Criteria:

* • All subjects aged 50y or more with recent fracture ankle (less than two weeks) with uncontrolled diabetes in form of high level of hemoglobinA1C ( >6.4% ) and/ or high random blood sugar level on admission (>200mg/dl). Patients with one or more complications due to diabetic e,g. neuropathy, nephropathy , and/or peripheral vascular disease.

Exclusion Criteria:

* • Previous ankle fracture fixation in the same side.

  * Charcot arthropathy
  * Polytrauma, multiple skeletal injury.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-09-30 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Complication rate | 6 months
  wound infection, hardware failure, Charcot arthropathy, development of ulcer

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt